CLINICAL TRIAL: NCT05895071
Title: Comparative Efficacy of Topical 5%Potassium Hydroxide vs Liquid Nitrogen in the Treatment of Plane Warts
Brief Title: Comparison of Topical 5%Potassium Hydroxide vs Liquid Nitrogen in the Treatment of Plane Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr sana aslam, Principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cmh abbottabad123
Record Dates: First submitted 2023-05-16; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Plan Warts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Topical 5% potassium hydroxide (Active Comparator): In group-A 30 patients were given topical 5%-potassium hydroxide solution on affected area once at night upto 4 weeks
  Interventions: Drug: 5%potassium hydroxide
- Group B Liquid nitrogen (Active Comparator): in group-B 30 patients treated with cotton bud method of cryotherapy with liquid nitrogen once every two weeks. Patients were reassessed at every two weeks and final assessment was done at 12th week.
  Interventions: Drug: Liquid nitrogen

INTERVENTIONS:
Drug: 5%potassium hydroxide — . In group-A 30 patients were given topical 5% potassium hydroxide solution on affected area once at night for upto 4 weeks
  Arms: Group A Topical 5% potassium hydroxide
Drug: Liquid nitrogen — in group-B 30 patients treated with cotton bud method of cryotherapy with liquid nitrogen once every two weeks. Patients were reassessed at every two weeks. The treatment carried out upto 12 weeks or until complete recovery from warts.
  Arms: Group B Liquid nitrogen

SUMMARY:
ABSTRACT Objective: To study the efficacy while comparing Potassium hydroxide 5% with liquid nitrogen in treatment of plane warts.

Study design: Randomized-controlled trial (RCT), (Double-blind). Study setting and duration: Dept dermatology, CMH-Abbottabad, Nov-2022 / April-2023.

Methodology: The sample size of 60 patients (children and adults aged 4 to 30 years) was calculated using Openepi app sample size RCT calculator, after informed consent by using non-probability consecutive sampling technique. Patients randomly assigned into two groups i.e. In group-A 30 patients were given topical 5%-potassium hydroxide solution on affected area once at night upto 4 weeks and in group-B 30 patients treated with cotton bud method of cryotherapy with liquid nitrogen once every two weeks. Patients were reassessed at every two weeks and final assessment was done at 12th week whereas followed up for 3 months to monitor recurrence. Demographic information and frequency percentages were calculated for qualitative variables by using SPSS26. To determine statistical significance taking p-value <0.05 as significant, and χ2-square test was used.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-30 years
* Both males and females
* Greater than 3 number of warts

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Those who are taking immunosupressive drugs

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Comparative Efficacy of topical 5% Potassium hydroxide and liquid nitrogen in the treatment of plane warts | 12 weeks
  Decrease in number or size of warts

CONTACTS AND LOCATIONS:
Locations (1):
- Sana aslam, Abbottabad, Khyber Pakhtun Khwaa, Pakistan